CLINICAL TRIAL: NCT02757898
Title: RBC Survival Validation in Adult Humans Under Condition of Normal RBC Survival
Brief Title: Transfusion of Biotinylated Red Blood Cells
Acronym: b-RBCs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, John D Roback, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00085954; R01HL095479-06 (NIH); P01HL086773-06A1 (NIH)
Record Dates: First submitted 2016-04-28; First posted 2016-05-02 (Estimated); Results first posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Anemia
Keywords: Red Blood Cell (RBC) transfusion; Biotin labeled red blood cells
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biotin-Labeled Red Blood Cell (RBC) Infusion (Experimental): Blood will be drawn from participants and labeled with biotin before being re-infused back to the participant. Blood samples will be obtained weekly over 10 weeks.
  Interventions: Drug: Biotin-Labeled Red Blood Cells (RBCs)

INTERVENTIONS:
Drug: Biotin-Labeled Red Blood Cells (RBCs) — 500 mL of blood will be drawn from each participant. The blood will be processed into a packed RBC unit.
  For participants 1 and 2, the RBCs will be labeled with biotin at three pre-defined concentrations of biotin labeling reagent (2, 6, 18 µg/mL of RBCs) and the labeled RBCs will be re-infused into the participant on the same day of collection.
  For participants 3 through 8, the RBCs will be stored at 2-6 C for 40-42 days before being labeled with three pre-defined concentrations of biotin labeling reagent (2, 6, 18 µg/mL of RBCs) and re-infused into the participant.
  Participants will have a 5 mL blood sample drawn within a few minutes of the re-infusion, the day after the re-infusion and then weekly for 70 days (10 weeks) to track the survival of the infused biotin labeled RBCs.

SUMMARY:
The purpose of this research is to study how red blood cells (RBCs) survive in a person's circulation, and how that survival may be different in red blood cells that are donated and stored prior to being transfused. Investigators will study this by collecting blood samples from participants, "labeling" RBCs with a naturally occurring vitamin, biotin. The RBCs will then be re-infused back into the participant and blood samples will be taken weekly for 10 weeks to assess the number of labeled cells in the samples.

DETAILED DESCRIPTION:
The purpose of this research is to study how red blood cells (RBCs) survive in a person's circulation, and how that survival may be different in red blood cells that are donated and stored prior to being transfused.

In this study, blood is collected from healthy subjects, processed into packed red blood cell units, and either immediately afterwards or 40-42 days later the packed red blood cells are labeled with biotin. The biotin-labeled red blood cells are then re-infused back to the donor (autologous transfusion). Blood samples are then taken from the subject every week for up to 70 days (10 weeks) to track survival of the labeled red blood cells.

This study also seeks to demonstrate that biotin-labeled RBCs can be safely transfused back to autologous subjects without any adverse reactions. All participants will be followed to watch for the development of antibodies against biotin-labeled RBCs.

ELIGIBILITY:
Inclusion Criteria:

* in good health

Exclusion Criteria:

* anemia (defined as hemoglobin < 8 g/dL)
* chronic disease, including diabetes, heart or lung disease, poorly managed hypertension, and peripheral vascular disease
* ongoing consumption of biotin or raw egg supplements
* history of a bleeding disorder
* evidence of anemia at initial screening
* women who are pregnant or plan to become pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2018-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D Roback, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Biotin-Labeled Red Blood Cell (RBC) Infusion: Blood will be drawn from participants and labeled with biotin before being re-infused back to the participant. Blood samples will be obtained weekly over 10 weeks.
  Biotin-Labeled Red Blood Cells (RBCs): 500 mL of blood will be drawn from each participant. The blood will be processed into a packed RBC unit.
  For participants 1 and 2, the RBCs will be labeled with biotin at three pre-defined concentrations of biotin labeling reagent (2, 6, 18 µg/mL of RBCs) and the labeled RBCs will be re-infused into the participant on the same day of collection.
  For participants enrolled after the first two participants, the RBCs will be stored at 2-6 C for 40-42 days before being labeled with three pre-defined concentrations of biotin labeling reagent (2, 6, 18 µg/mL of RBCs) and re-infused into the participant.
  Participants will have a 5 mL blood sample drawn within a few minutes of the re-infusion, the day after the re-infusion and then weekly for 70 days (10 weeks) to track the survival of the infused biotin labeled RBCs.
Period: Overall Study
Arm/Group | Biotin-Labeled Red Blood Cell (RBC) Infusion
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Biotin-Labeled Red Blood Cell (RBC) Infusion
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Had bRBC Detectable at 70 Days Post-intervention
Description: The length of time biotin-labeled RBCs can be detected following re-infusion. The number of participants was determined at day 70 by taking blood samples from each of them
Time Frame: 70 days post-intervention
Measure: Number; unit: participants
Groups:
- Biotin-Labeled Red Blood Cell (RBC) Infusion: Blood will be drawn from participants and labeled with biotin before being re-infused back to the participant. Blood samples will be obtained weekly over 10 weeks.
  Biotin-Labeled Red Blood Cells (RBCs): 500 mL of blood will be drawn from each participant. The blood will be processed into a packed RBC unit.
  For participants 1 and 2, the RBCs will be labeled with biotin at three pre-defined concentrations of biotin labeling reagent (2, 6, 18 µg/mL of RBCs) and the labeled RBCs will be re-infused into the participant on the same day of collection.
  For participants 3 through 5, the RBCs will be stored at 2-6 C for 40-42 days before being labeled with three pre-defined concentrations of biotin labeling reagent (2, 6, 18 µg/mL of RBCs) and re-infused into the participant.
  Participants will have a 5 mL blood sample drawn within a few minutes of the re-infusion, the day after the re-infusion and then weekly for 70 days (10 weeks) to track the survival of the infused biotin labeled RBCs.
Arm/Group | Biotin-Labeled Red Blood Cell (RBC) Infusion
Number analyzed (Participants) | 5
participants | 5

2. Primary Outcome: Length of Time Differentially Labeled Biotin-labeled RBCs Can be Distinguished From One Another
Description: The length of time that the three different concentrations of biotin labeling on the RBCs can be distinguished from one another will be determined by taking blood samples from each participant for 70 days
Time Frame: Up to 112 days
Population: For technical reasons, the investigators could not effectively label multiple red cell populations with different concentrations of biotin and this outcome was not collected.
Arm/Group | Biotin-Labeled Red Blood Cell (RBC) Infusion
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants Experiencing Adverse Events
Description: The total number of participants who experience adverse events, including development of anti-biotin-RBC antibodies will be determined. In previous studies, antibodies for biotin-labeled RBCs have been seen in a small number of people for up to 12 months.
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Biotin-Labeled Red Blood Cell (RBC) Infusion
Number analyzed (Participants) | 5
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 12 months after infusion.
Arm/Group | Biotin-Labeled Red Blood Cell (RBC) Infusion
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/98/NCT02757898/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT02757898/ICF_001.pdf